CLINICAL TRIAL: NCT05225753
Title: Post-operative Anemia in Lateral Fragility Fractures of the Femur. A Prospective Observational Study in Three Different Intramedullary Nails
Brief Title: Post-operative Anemia in Lateral Fractures of the Femur.
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: Ospedali Riuniti di Foggia (Other)
Responsible Party: Sponsor
Other Study IDs: Post-op Anemia
Record Dates: First submitted 2022-01-19; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2021-12

CONDITIONS: Femur Fracture
Keywords: fragility lateral femoral fractures; intramedullary nail; Post-operative anemia; surgical time; Blood transfusions number
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients treated with Affixus Zimmer-Biomet
  Interventions: Diagnostic Test: hemoglobin serum value
- patients treated with EBA2 Citieffe
  Interventions: Diagnostic Test: hemoglobin serum value
- patients treated with Proximal Femoral Nail Antirotation Synthes
  Interventions: Diagnostic Test: hemoglobin serum value

INTERVENTIONS:
Diagnostic Test: hemoglobin serum value — post-operative anemia evaluated with hemoglobin serum value

SUMMARY:
It was conducted a prospective study with a series of 45 patients with lateral fragility fractures of the femur treated by three different intramedullary nails. Patients were randomized in Group A (15 patients treated by Affixus Zimmer-Biomet), Group B (15 patients treated by EBA2 - Citieffe) and Group C (15 patients treated by Proximal Femoral Nail Antirotation Synthes).

One independent observer performed seven biochemical evaluations (hemoglobin serum value) from admission to patient discharge. Surgical time and Blood transfusions number were reported for each partecipant.

ELIGIBILITY:
Inclusion Criteria:

* femur fractures type 31-A1, A2, A3 (Muller ME, Nazarian S, Kock P et al.);
* age more than 65 years;

Exclusion Criteria:

* patients with neurological diseases;
* finding of anemia before surgery;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Fortyfive (45) patients referring to the Orthopaedic and Trauma Unit of the local University Hospital between November 2020 and September 2021 with lateral fragility fracture were prospectively recruited.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin serum value | Preoperative, Day 0, Day 1, Day 2, Day 3, Day 5 (after surgery)
  Post-operative anemia was quantified using the hemoglobin serum value ranging between more than 10 g/dl (no post-operative anemia) and less than 10 g/dl (post-operative anemia).

CONTACTS AND LOCATIONS:
Locations (1):
- AOUC Policlinico di Bari - UOC Ortopedia e Traumatologia, Bari, Italy